CLINICAL TRIAL: NCT03049501
Title: A Tailored Technology Intervention for Diverse Caregivers of AD Patients
Brief Title: Caring for the Caregiver Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, David Loewenstein, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20130460; R01NR014434 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Caregivers of Alzheimer's Disease or Memory Problem Patients
Keywords: Alzheimer's caregivers; Technology-based intervention; Culturally-tailored intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiving Condition (Experimental): Participants will receive a computer tablet and have access to web-based skill building sessions, videos from experts, annotated resources and information and tips on caregiving-related topics
  Interventions: Behavioral: Caregiving condition
- Nutrition Condition (Placebo Comparator): Participants will receive a computer tablet and have access to web-based training sessions on different topics related to nutrition.
  Interventions: Behavioral: Nutrition condition

INTERVENTIONS:
Behavioral: Caregiving condition — The intervention will consist of multimedia features accessible via the study-provided tablet. The components include: skill-building sessions and modules; a resource guide; an annotated reading list; information and tips; expert educational seminars (video); and structured support group sessions (6 sessions). All the sessions (home-based, one-on-one, and support group sessions) will last about 60-90 minutes.
  Arms: Caregiving Condition
Behavioral: Nutrition condition — The intervention will provide resource and information tips on topics related to Nutrition for a total of 8 sessions. The first and last session will be home-based and all the other sessions will be conducted via web-conferencing using the tablet provided.
  Arms: Nutrition Condition

SUMMARY:
The prevalence of family caregivers is projected to increase in concert with the projected increase in number of AD patients. The focus of the study is to gather systematic data on the acceptability and efficacy of a unique technology-based, culturally- tailored psycho-social intervention program that targets ethnically/culturally diverse family caregivers of patients with Alzheimer's Disease. The overall goal of the project is to improve the lives of family caregivers as well as their ability to provide care to their loved one and to reduce disparities in access to needed services and support among caregiver populations.

ELIGIBILITY:
Inclusion Criteria:

1. Speak and understand English or Spanish
2. Provide care to a loved one with memory decline
3. Not having terminal illness/condition
4. 18+ yrs old

Exclusion Criteria:

1. Not providing care to a loved one with Alzheimer disease or dementia
2. Not speak English or Spanish
3. Have cognitive deficit
4. Have terminal illness
5. Plan to place their loved one in a facility
6. Plan to move away in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2013-07; Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Loewenstein, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregiving Condition: Participants will receive a computer tablet and have access to web-based skill building sessions, videos from experts, annotated resources and information and tips on caregiving-related topics
  Caregiving condition
- Nutrition Condition: Participants will receive a computer tablet and have access to web-based training sessions on different topics related to nutrition
  Nutrition condition
Period: Overall Study
Arm/Group | Caregiving Condition | Nutrition Condition
Started | 123 | 121
6 Month Follow up | 107 | 91
12 Month Follow up | 101 | 92
Completed | 101 | 92
Not Completed | 22 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiving Condition | Nutrition Condition | Total
Number analyzed (Participants) | 123 | 121 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 82 | 150
  >=65 years | 55 | 39 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 101 | 204
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 54 | 109
  Not Hispanic or Latino | 68 | 67 | 135
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 26 | 55
  White | 85 | 89 | 174
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Depression as Measured by Center for Epidemiologic Studies Depression Scale (CES-D)
Description: CES-D Scale ranges from 0 to 30 with higher scores indicating greater frequency of depressive symptoms.
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: Follow up visits were not completed for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving Condition | Nutrition Condition
Number analyzed (Participants) | 123 | 121
score on a scale
  Baseline | 11.38 (7.02) | 10.88 (5.79)
  6 month follow up: number analyzed (Participants) | 107 | 91
  6 month follow up | 10.86 (6.63) | 10.69 (6.23)
  12 month follow up: number analyzed (Participants) | 101 | 92
  12 month follow up | 10.32 (7.18) | 10.46 (6.25)

2. Primary Outcome: Caregiving Burden as Measured by Burden Inventory
Description: Higher score means greater level of caregiver burden. Range (0-44)
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: Follow up visits were not completed for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving Condition | Nutrition Condition
Number analyzed (Participants) | 123 | 121
score on a scale
  Baseline | 18.52 (8.91) | 19.66 (7.59)
  6 month follow up: number analyzed (Participants) | 107 | 91
  6 month follow up | 16.89 (8.39) | 18.23 (6.97)
  12 month follow up: number analyzed (Participants) | 101 | 92
  12 month follow up | 16.08 (8.29) | 17.66 (8.27)

3. Primary Outcome: Caregiver's Self Report of Self-care
Description: A 13 Item self care questionnaire is used to measure caregivers self care. Each item can be scored as 0,1,negative 3 or negative 4. The total score ranging from negative 52 to 13. Higher score means better in keeping medical obligations to him/herself.
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: Follow up visits were not completed for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving Condition | Nutrition Condition
Number analyzed (Participants) | 123 | 121
score on a scale
  Baseline | 0.62 (0.18) | 0.60 (0.17)
  6 month follow up: number analyzed (Participants) | 107 | 91
  6 month follow up | 0.62 (0.18) | 0.60 (0.17)
  12 month follow up: number analyzed (Participants) | 101 | 92
  12 month follow up | 0.62 (0.20) | 0.61 (0.17)

4. Primary Outcome: Caregiver's Self-report of Physical Health
Description: SF 12 Health Survey was used to measure physical health of the caregiver. Scores ranges from 0 to 35 with lower score means less limitation to physical health.
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: Follow up visits were not completed for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving Condition | Nutrition Condition
Number analyzed (Participants) | 123 | 121
score on a scale
  Baseline | 2.71 (1.03) | 2.75 (1.14)
  6 month follow up: number analyzed (Participants) | 107 | 91
  6 month follow up | 2.89 (1.12) | 2.51 (1.11)
  12 month follow up: number analyzed (Participants) | 101 | 92
  12 month follow up | 2.76 (1.09) | 2.67 (1.22)

5. Primary Outcome: Caregiver's Self-efficacy
Description: A 15 item Caregiver's self efficacy questionnaire will be used to assess caregiver's self-efficacy. The questionnaire score ranges from 0-1500 percent with a lower percentage score indicating less efficacy.
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: Follow up visits were not completed for all participants
Measure: Mean (Standard Deviation); unit: percentage of efficacy
Arm/Group | Caregiving Condition | Nutrition Condition
Number analyzed (Participants) | 123 | 121
percentage of efficacy
  Baseline | 925.21 (243.36) | 936.65 (249.62)
  6 month follow up: number analyzed (Participants) | 107 | 91
  6 month follow up | 971.43 (295.41) | 964.15 (273.06)
  12 month follow up: number analyzed (Participants) | 101 | 92
  12 month follow up | 999.65 (285.94) | 1047.71 (225.14)

6. Primary Outcome: Positive Aspects of Caregiving
Description: An 11 item positive aspects of caregiving questionnaire was used to measure positive aspects of caregiving. Each item can be scored 0, 1, 2, 3, 4, negative 3 or negative 4. The total score ranging from negative 44 to 44. Higher score means more positive feelings towards caregiving.
Time Frame: Baseline, 6-mth follow-up and 12-mth follow-up
Population: Follow up visits were not completed for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving Condition | Nutrition Condition
Number analyzed (Participants) | 123 | 121
score on a scale
  Baseline | 24.46 (8.49) | 23.24 (8.83)
  6 month follow up: number analyzed (Participants) | 107 | 91
  6 month follow up | 24.72 (8.34) | 24.02 (8.54)
  12 month follow up: number analyzed (Participants) | 101 | 92
  12 month follow up | 24.00 (9.60) | 24.58 (8.54)

ADVERSE EVENTS:
Description: Per protocol, adverse events will not be collected during the course of this study.
Arm/Group | Caregiving Condition | Nutrition Condition
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT03049501/Prot_SAP_000.pdf